CLINICAL TRIAL: NCT00690144
Title: Prospective Study Focusing on Impact of High-fidelity Simulation in Health Care Education
Brief Title: High-fidelity Simulation in Health Care Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Matthew Huei-Ming Ma, MD, PhD, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 200803078R
Record Dates: First submitted 2008-05-28; First posted 2008-06-04 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: simulation; medical education; performance of clinical reasoning and skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- simulation group (Experimental): the trainees in the simulation group receive simulation-based training
  Interventions: Device: High-fidelity high-fidelity mannequin simulator (SimMan, Laerdal, Stavanger, Norway).

INTERVENTIONS:
Device: High-fidelity high-fidelity mannequin simulator (SimMan, Laerdal, Stavanger, Norway). — Critical care training using high-fidelity simulation. The case scenarios were simulated by a high-fidelity mannequin simulator (SimMan, Laerdal, Stavanger, Norway).

SUMMARY:
The purpose of this study is to determine whether the use of high-fidelity simulation in health care education is an effective training and evaluation model.

DETAILED DESCRIPTION:
High-fidelity simulation has many advantages in medical education. Simulation-based critical care training is especially valuable due to error-prone work settings and the high cost of patient adverse events. This study was conducted to assess the effectiveness of implementing the high-fidelity simulation in critical care training, and the feasibility of high-fidelity simulation as an evaluation tool.

ELIGIBILITY:
Inclusion Criteria:

* healthcare trainees, including medical students, nursing students, residents, nursing staff and emergency medical technicians.

Exclusion Criteria:

* any trainees unwilling to receive simulation-based training

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2007-07; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
performance of clinical reasoning and skills in simulated settings | before and after the simulation-based training

SECONDARY OUTCOMES:
clinical performance of reasoning and skills | before and after the simulation-based training

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Huei-Ming Ma, MD, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan